CLINICAL TRIAL: NCT03119025
Title: Safety/Efficacy of Vaccination With Autologous Dendritic Cells Pulsed With Recombinant HCV-Antigens (Core and NS3) for Treatment of Patients With Chronic HCV-Infection
Brief Title: Autologous Dendritic Cell Vaccine for Treatment of Patients With Chronic HCV-Infection
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Russian Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Alexander A Ostanin, Head of Clinical Department, Russian Academy of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IFCI-04/10/2015
Record Dates: First submitted 2017-03-27; First posted 2017-04-18 (Actual); Results first posted 2019-05-10 (Actual); Last update posted 2019-05-10 (Actual); Status verified 2019-02

CONDITIONS: Hepatitis C, Chronic; Liver Diseases; Hepatitis; Virus Diseases
Keywords: Dendritic Cells; DC-based Vaccines; Chronic HCV Infection; Antigen-Specific T cell response; Recombinant HCV-Core antigen; Recombinant HCV-NS3 antigen
MeSH Terms: conditions — Hepatitis C, Chronic; Liver Diseases; Hepatitis; Virus Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Autologous DC-vaccines (Experimental): Thirty patients with chronic hepatitis C (genotype 1) will receive the initiating and maintaining courses of autologous of autologous monocyte-derived dendritic cells, generated in the presence of IFN-α/GM-CSF and pulsed with recombinant HCV Core (1-120) and NS3 (1192-1457) proteins.
  Interventions: Biological: Autologous DC-vaccines

INTERVENTIONS:
Biological: Autologous DC-vaccines — Patients will be vaccinated via intracutaneous injection of autologous DCs (5×106) combined with adjuvant subcutaneous injection of recombinant hIL-2 (250 000 IU).
  Initiating course: one vaccination per week, during 1 month. Maintaining course: one vaccination per month, during 6 month. Patients will be monitored in a 2 months (after completing of initiating course), 7 months (after completing of maintaining course) and 13 months (in a 6 months post-vaccination follow-up).

SUMMARY:
Clearance of HCV infection requires early and multi-specific HLA class I restricted CD8+ T cell and class II restricted CD4+ T cell responses to both structural (Core) and non-structural HCV proteins (NS3, NS4A, NS5A, NS5B). Dendritic cells (DCs) are professional antigen-presenting cells that link innate and adaptive immune responses, and play a major role in priming, initiating, and sustaining strong anti-HCV T cell immune responses.

The general objective of this study is to evaluate safety, feasibility and clinical efficacy of therapeutic vaccination in genotype 1 HCV patients using autologous DCs pulsed with recombinant HCV-antigens (Core and NS3). Expected effects: DC vaccination induces Core/NS3-specific immune response and reduces viral load in patients with chronic HCV-infection.

DETAILED DESCRIPTION:
Hepatitis C virus (HCV) has chronically infected an estimated 170 million people worldwide. People infected with HCV are at risk for developing chronic liver diseases, such as liver cirrhosis and primary hepatocellular carcinoma. It has been estimated that HCV accounts for 27% of cirrhosis and 25% of hepatocellular carcinoma worldwide. Therapy for chronically HCV-infected patients has involved a pegylated interferon-alpha and ribavirin (pegIFN/RBV) and is still the only FDA-approved therapeutic combination. However, this therapy is expensive, non-specific, toxic, and only effective in about 50% of genotype-1 HCV patients.

An early immune response, represented by the activation of NK cells, the development of vigorous anti-HCV CD4+ and CD8+ T-cell responses, and the appearance of HCV-specific antibodies, is mounted by the host during acute HCV infection and leads to clearance of the virus. However, in the vast majority (≈85%) of infected individuals HCV causes a persistent infection. The mechanisms of HCV persistence remain elusive and are largely related to inefficient clearance of the virus by the host immune system.

Although HCV genome is very variable with hundreds of serotypes and six genotypes, several structural (Core) and nonstructural proteins (NS3, NS4A, NS5A, NS5B) are highly conserved among genotypes and subtypes. It is apparent that clearance of hepatitis C infection requires early and multi-specific HLA class I restricted CD8+ T cell and class II restricted CD4+ T cell responses to both structural and non-structural HCV proteins.

DCs are professional antigen-presenting cells that link innate and adaptive immune responses. DCs play a major role in priming, initiating, and sustaining strong T cell responses against pathogen-derived antigens. Therefore DC-based therapy represents a promising immunotherapeutic approach in terms of their propensity to establish anti-HCV adaptive immune responses.

This trial is a prospective, non-blinded, interventional study to determine safety, feasibility and clinical efficacy of therapeutic vaccination in genotype 1 HCV patients using autologous DCs pulsed with recombinant HCV-antigens (Core and NS3). Our previous work has shown that the short-term loading of DCs with recombinant HCV proteins Core (1-120) and NS3 (1192-1457) have no any marked inhibitory effect on maturation and functions of DCs.

In experimental group thirty patients with chronic hepatitis C (genotype 1) will be vaccinated via intracutaneous injection of monocyte-derived DCs, generated in the presence of IFN-α/GM-CSF and pulsed with recombinant HCV Core (1-120) and NS3 (1192-1457) proteins. The vaccination protocol will includes initiating (one injection per week, no 4) and maintaining (one injection per month, no 6) courses with subsequent 6-month of follow up.

The safety will be determined by the evaluation of the number of participants with the adverse events. Liver safety will be assessed by blood analysis and Ultrasound. Patients will be monitored in a 2 months (after completing of initiating course), 7 months (after completing of maintaining course) and 13 months (in a 6 months post-vaccination follow-up).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 65 Years (Adult)
* Chronic hepatitis C (genotype 1b)
* HCV-positive patients
* Plasma HCV RNA level ≥ 10 000 IU/ml
* Liver fibrosis (METAVIR Score 0-III)
* Patients must be able to tolerate all study procedures
* Patients must be willing to voluntarily give written Informed Consent to participate in the study before any procedures are performed
* Patients must be willing to be available for all baseline, treatment and follow-up examinations required by protocol

Exclusion Criteria:

* Co-infection with hepatitis B, A, D, E, cytomegalovirus or Epstein-Barr virus
* Liver cirrhosis (METAVIR Score IV)
* The high degree of hepatitis activity (ALT and/or AST ≥ 10 ULN)
* Received any vaccine within a month prior to study entry
* A history of diabetes
* Psychiatric disorders
* Renal dysfunctions
* Hemodynamic or respiratory instability
* HIV or uncontrolled bacterial, fungal, or viral infections
* Autoimmune diseases
* Pregnancy
* Malignancy
* Participation in other clinical trials

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elena R Chernykh, MD, PhD, Study Chair — Institute of Fundamental and Clinical Immunology; Alexander A Ostanin, MD, PhD, Principal Investigator — Institute of Fundamental and Clinical Immunology
Locations (1):
- Institute of Fundamental and Clinical Immunology, Novosibirsk, Russia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Oleynik EA, Leplina OY, Tyrinova TV, Tikhonova MA, Pyrinova GB, Ostanin AA, Starostina NM, Chernykh ER. The influence of recombinant HCV proteins Core and NS3 on maturation and functions of dendritic cells generated in vitro with interferon-alpha. Immunology 37 (5): 239-245, 2016. (in Russian) DOI: 10.18821/0206-4952-2016-37-5-239-245
- Available data/document: Clinical Study Report — https://doi.org/10.1007/s12026-017-8967-2 — Chernykh E., Leplina O., Oleynik E., Tikhonova M., Tyrinova T., Starostina N., Ostanin A. Immunotherapy with interferon-α-induced dendritic cells for chronic HCV infection (the results of pilot clinical trial) // Immunologic Research.- 2017

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment, assessment and treatment of patients were conducted from May 2015 to November 2016 in a Clinic of Immunopathology affiliated with Institute of Fundamental and Clinical Immunology, that currently holds a license for cell technology application.
Groups:
- Autologous DC-vaccines: Ten patients with chronic hepatitis C (genotype 1) were received the initiating and maintaining courses of autologous monocyte-derived dendritic cells, generated in the presence of IFN-α/GM-CSF and loaded with recombinant HCV Core (1-120) and NS3 (1192-1457) proteins.
  Autologous DC-vaccines: Patients were vaccinated via intracutaneous injection of autologous DCs (5×106) combined with adjuvant subcutaneous injection of recombinant hIL-2 (250 000 IU).
  Initiating course: one vaccination per week, during 1 month. Maintaining course: one vaccination per month, during 6 month. Patients were monitored at baseline (before the first vaccination) and in a 2 months (after completing of initiating course), 7 months (after completing of maintaining course) and 13 months (in a 6 months post-vaccination follow-up).
Period: Overall Study
Arm/Group | Autologous DC-vaccines
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Autologous DC-vaccines
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 35.5 [31 to 45]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Russia | 10
Patients with chronic hepatitis C (genotype 1b) [Count of Participants; unit: Participants] | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Severe Adverse Reactions and/or With Abnormal Clinical Laboratory Values That Are Related to Treatment
Description: Frequency of severe adverse reactions will be evaluated from enrollment and up to 13 months. Liver safety by blood analysis (ALT, AST, GGT, Total and conjugated bilirubin, platelets, ESR, etc) and Ultrasound will be assessed from enrollment and up to 13 months (= baseline, 2, 7 and 13 months after 1-st vaccination).
Time Frame: From enrollment and up to 13 months
Population: Most patients had minimal hepatitis activity as evidenced by normal or slightly increased liver transaminase levels. Serum HCV RNA levels ranged from 1.3 × 104 IU/mL to 1.8 × 106 IU/mL. Fibrosis stage ranged from F0 to F3 according to Metavir system scores.
Measure: Count of Participants; unit: Participants
Groups:
- Autologous DC-vaccines: Ten patients with chronic hepatitis C (genotype 1) were received the initiating and maintaining courses of autologous of autologous monocyte-derived dendritic cells, generated in the presence of IFN-α/GM-CSF and loaded with recombinant HCV Core (1-120) and NS3 (1192-1457) proteins.
  Autologous DC-vaccines: Patients were vaccinated via subcutaneous injection of autologous DCs (5×106) combined with adjuvant subcutaneous injection of recombinant hIL-2 (250 000 IU).
  Initiating course: one vaccination per week, during 1 month. Maintaining course: one vaccination per month, during 6 month. Patients were monitored at baseline (before the first vaccination) and in a 2 months (after completing of initiating course), 7 months (after completing of maintaining course) and 13 months (in a 6 months post-vaccination follow-up).
Arm/Group | Autologous DC-vaccines
Number analyzed (Participants) | 10
Participants | 0

2. Secondary Outcome: Number of Participants With Virological Response According to HCV RNA Viral Load
Description: Virological response in patients receiving DC-vaccinations is defined as change from baseline in HCV RNA viral load by at least 1 log at 2, 7 and 13 month after 1-st vaccination. Plasma level of HCV RNA will be measured by Real-Time Reverse Transcription-Polymerase Chain Reaction (RT-PCR)
Time Frame: Baseline, 2, 7 and 13 months after 1-st vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | Autologous DC-vaccines
Number analyzed (Participants) | 10
Participants | 4

3. Secondary Outcome: Number of Participants Who Have Developed or Increased Anti-Viral Immune Response According to T-cell Proliferation
Description: Change from baseline in T-cell proliferative response to HCV Core and NS3 proteins at 2, 7 and 13 month after 1-st vaccination. T-cell proliferation will be evaluated using radiometry based on 3H-thymidine incorporation
Time Frame: Baseline, 2, 7, and 13 months after 1-st vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | Autologous DC-vaccines
Number analyzed (Participants) | 10
Participants | 9

4. Secondary Outcome: Number of Participants Who Have Developed or Increased Anti-Viral Immune Response According to IFN-γ Production
Description: Change from baseline in T-cell IFN-γ-producing response to HCV Core and NS3 proteins at 2, 7 and 13 month after 1-st vaccination. Production of IFN-γ will be measured by ELISA kit
Time Frame: Baseline, 2, 7 and 13 months after 1-st vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | Autologous DC-vaccines
Number analyzed (Participants) | 10
Participants | 9

ADVERSE EVENTS:
Time Frame: Frequency of adverse events was evaluated from enrollment and up to the end of 13 months.
Description: The number of participants with Adverse Events was zero because i) patients had minimal hepatitis activity without severe concomitant diseases or bacterial/fungal/virus co-infections; ii) patients were received autologous (not allogenic or xenogenic) DCs in low doses (5 × 106/vaccination) via intracutaneous (not intravenous or intrahepatic) injections and adjuvant subcutaneous injection of rhIL-2 (Roncoleukin - Russian pharmaceutical product) in minimal doses (250 000 IU).
Arm/Group | Autologous DC-vaccines
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2015-04-10): https://cdn.clinicaltrials.gov/large-docs/25/NCT03119025/Prot_000.pdf
  • Statistical Analysis Plan (2015-04-10): https://cdn.clinicaltrials.gov/large-docs/25/NCT03119025/SAP_001.pdf
  • Informed Consent Form (2015-04-10): https://cdn.clinicaltrials.gov/large-docs/25/NCT03119025/ICF_002.pdf